CLINICAL TRIAL: NCT05922566
Title: The Exploration of the Effect of Mukbang on Functional Connectivity of Related Brain Regions in Children With Cancer Hospitalized for Radiotherapy and Chemotherapy Based on fMRI
Brief Title: Research on the Influence of Mukbang on Brain Activation in Children With Cancer Based on fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: fMRI
Record Dates: First submitted 2023-05-22; First posted 2023-06-28 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Children With Cancer
Keywords: childhood cancer; Mukbang; Functional magnetic resonance imaging; appetite
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fMRI scanning while Mukbang watching (Experimental): The fMRI scanning will be divided into 3 parts, includes structural image scans, resting state scans, and task state scans. For the task state function image scanning, participants will be asked to watch the specific video program which includes the food images and eating sound of Mukbang and General short videos without food cues.
  Healthy kids and children with cancer hospitalized for radiotherapy and chemotherapy will both accept this intervention.
  Interventions: Combination Product: fMRI + Mukbang videos

INTERVENTIONS:
Combination Product: fMRI + Mukbang videos — Specific video program + fMRI will be allocated to the participants in this group. The specific video program includes control videos without food information, eating and food images without sound, chewing and swallowing sound without images, and Interactive content in Mukbang. Participants will undergo structural image scans, resting state scans, and task state scans. The task-fMRI will be performed while watching Mukbang to explore the activation of brain functional areas.

SUMMARY:
This study aims to use the intervention study method to extract and verify the effective ingredients in Mukbang that promote appetite and eating in children with tumor during radiotherapy and chemotherapy, and to analyze and explore their potential mechanisms of action based on functional magnetic resonance imaging.

DETAILED DESCRIPTION:
Cancer has a high incidence among children and adolescents worldwide. In October 2020, the World Health Organization (WHO) released an overview of the Global Action on Childhood Cancer which showed that more than 400,000 children under the age of 19 were diagnosed with cancer worldwide every year. With the development and progress of diagnosis and treatment technology, the health outcome of children with cancer has been greatly improved.

However, the side effects and complications associated with cancer and its treatment can seriously affect the appetite and food intake of children with cancer, resulting in malnutrition and a low quality of life. Therefore, it is very important to effectively improve the appetite of children with cancer during treatment.

Clinical methods to improve the appetite of cancer patients mainly include drugs, diet or nutrition intervention, traditional Chinese medicine and acupuncture, but each intervention has its own advantages and disadvantages which makes the clinical application effect difficult to evaluate, in urgent need of more effective solutions to solve this problem.

Mukbang has shown great potential in helping children with cancer to improve their appetite and food consumption, finally promote nutritional health. Mukbang is a method independently chosen by hospitalized cancer children with radiotherapy and chemotherapy to help promote appetite, which has a natural high acceptance. What's more, the features of Mukbang, such as high-quality and clear pictures, relaxed atmosphere created by the video makers, sounds while eating, and attractive images of food, may promote viewers' appetite and increase their intake imperceptibly.

In addition to that, watching Mukbang while eating can also provide a pleasant eating experience for children with cancer, and the interaction with the Mukbang anchor can also alleviate the loneliness of children who live in hospital for such a long time, so as to enhance the children's taste experience, relieve the negative emotions of loneliness and depression and promote their appetite and interest in food under the condition of ensuring a healthy diet.

Research has found that Mukbang can help people with low appetites increase their food intake and provide vicarious satisfaction to those who overeat. Several studies have shown that videos containing food cues can increase viewers' appetite and decrease feelings of satiety to a certain extent. At the same time, Mukbang can also increase viewers' taste experience on the basis of physics and improve children's interest in food.

Therefore, on the basis of existing studies, this study will use functional magnetic resonance imaging and cross-case analysis to extract and verify the effective ingredients in Mukbang that promote appetite and eating in children with tumor during radiotherapy and chemotherapy, and analyze and discuss their potential mechanism of action, aiming to provide a new direction for clinical departments to develop nutritional intervention measures and management programs for children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* children with cancer aged between 10 to 18 years old;
* diagnosed with any tumor or cancer other than brain tumor before the age of 18;
* having received or are receiving inpatient treatment;
* both the patient and the guardian can communicate in Chinese;
* children with moderate or higher symptoms of decreased appetite were screened for the Therapy-Related Symptom Checklist for Children.

Exclusion Criteria:

* a diagnosis of a serious disease other than a tumor, especially a brain disease such as epilepsy and organic psychosis, was identified from the case;
* unable to complete communication due to serious mental or physical illness, such as cognitive impairment or unclear consciousness;
* children with eye or ear dysfunction that prevents them from watching and listening to videos;
* with braces, cardiac pacemakers and other items with iron magnetism that cannot be removed from the body;
* people who suffer from claustrophobia, ADHD, and other problems of staying quiet in confined spaces for long periods of time.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The pictures of activated functional areas of the brain | Baseline
  The outcome can be collected using the Siemens 3T Prisma functional Magnetic Resonance Imaging machine with an Inspur data processing system. The pictures reflect the brain functional areas which can be activated by watching Mukbang.

SECONDARY OUTCOMES:
Cancer Appetite and Symptom Questionnaire, CASQ | Change from baseline appetite at 1 hour intervention
  Participants' self-reported appetite, to reflect the participants' own perceived appetite.
The number of increased salivation and perceived appetite | Change from baseline salivation and perceived appetite during 1 hour fMRI scanning
  In order to further evaluate the relationship between the functional activities of the appetition-related regions of the brain and appetite, the number of salivation and increased perceived appetite will be recorded by pressing the button during the MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.